CLINICAL TRIAL: NCT06820255
Title: Prospective Evaluation of the DDR Genes Alteration to Predict Response to Platinum-based Chemotherapy in Advanced Urothelial Cancer.
Brief Title: DDR Genes Alteration and Response to Platinum-based Chemotherapy in Advanced Urothelial Cancer.
Acronym: SELECTIO-UC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 7004; 2024-516450-21 (EudraCT Number)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer Metastatic or Unresectable; Upper Tract Urothelial Cancer
Keywords: DNA damage response genes; cisplatin; carboplatin
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Platinum; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Patients will be screened for DDR alteration on tumor tissue and treated with platinum-based chemotherapy followed by avelumab maintenance.
  Outcome to therapy will be evaluated based on presence or not of DDR alterations.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both patients and clinicians are blinded for results of DDR test during platinum-based chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DDR alterations positive (Active Comparator): This arm included all patients with DDR alteration in urothelial cancer
  Interventions: Drug: Platinum + Gemcitabine; Drug: Avelumab first-line maintenance; Diagnostic Test: NGS test for DDR alterations
- DDR alterations negative (Active Comparator): This arm included all patients without DDR alteration in urothelial cancer
  Interventions: Drug: Platinum + Gemcitabine; Drug: Avelumab first-line maintenance; Diagnostic Test: NGS test for DDR alterations

INTERVENTIONS:
Drug: Platinum + Gemcitabine — Eligible patients will be treated with platinum-based chemotherapy (i.e. cisplatin + gemcitabine or carboplatin + gemcitabine).
Drug: Avelumab first-line maintenance — Patients with stable disease or tumor response after treatment with platinum-based chemotherapy will start treatment with avelumab 800 mg fat dose Q2 weeks until progression of disease or unacceptable toxicity
Diagnostic Test: NGS test for DDR alterations — All patients will be tested for DDR alterations on tumor tissue.

SUMMARY:
This study aims to prospectively observe whether certain alterations in some genes related to the DNA repair mechanism are related to better response to platinum-based chemotherapy used to treat metastatic bladder or urothelial cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-specific procedures. Patients must be able to understand and be willing to sign a written informed consent.
2. Male or female patient ≥18 years of age.
3. Histological or cytological documentation of urothelial cancer.
4. Available tumor tissue for analysis
5. Measurable disease according to Response Evaluation Criteria in Solid Tumors criteria, version 1.1.
6. Eastern Cooperative Oncology Group performance status of ≤2. (Patients with ECOG PS of 2 were required to also meet the additional criteria: hemoglobin ≥10 g/dL, GFR ≥50mL/min, may not have NYHA class III heart failure).
7. Life expectancy of at least 6 months.
8. Eligible to standard chemotherapy with cisplatin or carboplatin + gemcitabine as per clinical practice.
9. Women of childbearing potential and men must agree to use adequate contraception since signing of the informed consent form until 180 days after the last dose of chemotherapy and 30 days after the last dose of avelumab. The investigator or a designated associate is requested to advise the subject how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommend method (or combination of methods) as per standard of care.
10. Adequate bone-marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days of starting to study treatment:

a Creatinine value <2.5 mg/dl and creatinine clearance > 30 ml/min evaluated by the Cockcroft-Gault Formula.

b Total bilirubin ≤1∙5 × the upper limit of normal (ULN); c Alanine aminotransferase and aspartate aminotransferase ≤2 × ULN (≤5 × ULN for patients with liver involvement of their cancer); d International normalized ratio (INR) and partial thromboplastin time (PTT) ≤1∙5 × ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no prior evidence of an underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care; e Platelet count ≥100 000/mm3, hemoglobin >9 g/dl, absolute neutrophil count >1,500/mm3; f Alkaline phosphatase limit ≤2∙5 × ULN (≤5 × ULN for patients with liver involvement of their cancer).

Exclusion Criteria:

1. Previous treatment for metastatic or locally advanced disease.
2. Previous adjuvant therapy within 1 year from the diagnosis of metastatic disease.
3. Prior treatment with immunotherapy.
4. Previous or concurrent cancer that is distinct in primary site or histology from urothelial cancer within 3 years before enrollment EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors (Ta [non-invasive tumor], Tis [carcinoma in situ], and T1 [tumor invades lamina propria]), pT2 prostate cancer with PSA<0.01.
5. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
6. Pregnancy or breast-feeding. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.
7. Any cardiological condition among:

   1. Congestive heart failure of New York Heart Association class 3 or worse.
   2. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of study drug.
   3. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted).
   4. Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management).
   5. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), pulmonary embolism within the 4 months before start of study medication.
8. Ongoing infection higher than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 grade 2.
9. Known history of human immunodeficiency (HIV) virus infection or known history of chronic hepatitis B or C.
10. Any autoimmune disease that contraindicates the use of maintenance immunotherapy in case of stable or responsive disease to chemotherapy.
11. Seizure disorder requiring medication.
12. Symptomatic metastatic brain or meningeal tumors unless the patient is >2 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. Also, the patient must not be undergoing acute steroid therapy or tapering (chronic steroid therapy is acceptable provided that the dose is stable for 1 month before and after screening radiographic studies).
13. History of organ allograft.
14. Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event of CTCAE grade 3 or higher within 4 weeks of start of study medication.
15. Non-healing wound, ulcer, or bone fracture.
16. Renal failure requiring hemodialysis or peritoneal dialysis.
17. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his or her compliance in the study.
18. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
19. Participation to another clinical trial at the time of the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by DDR group. | Six months
  The difference in ORR defined as the percentage of patients who achieve PR or CR as measured by RECIST 1.1, to the platinum-based chemotherapy between patients with metastatic or locally advanced urothelial cancer with or without DDR genes alterations.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by DDR group. | 12 months
  The PFS defined as the time elapsed from start of investigational treatment to the documentation of investigator-assessed disease progression, according to RECIST 1.1 [22], or death due to any cause, whichever occurs first in patients with or without DDR genes alterations.
Overall Survival (OS) by DDR group. | 12 months
  The OS is defined as time elapsed from start of treatment to the date of death due to any cause in patients with or without DDR genes alterations.
Overall Response Rate (ORR) by treatment group. | six months
  The ORR is defined as the percentage of patients who achieve PR or CR as measured by RECIST 1.1 criteria in patients with or without DDR genes alterations between those treated with carboplatin o cisplatin.
Disease Control Rate (DCR) by treatment group. | six months
  The disease control rate (DCR) is defined as the percentage of patients who achieve stable disease (SD), or PR or CR as measured by RECIST 1.1 criteria in patients treated with carboplatin o cisplatin.
Disease Control Rate (DCR) by DDR group. | six months
  The disease control rate (DCR) is defined as the percentage of patients who achieve stable disease (SD), or PR or CR as measured by RECIST 1.1 criteria in patients with or without DDR genes alterations.
Treatment-related toxicity | 12 months.
  The treatment-related toxicity will be evaluated by the incidence of chemo-related adverse events in patients with or without DDR genes alterations graded according to NCI CTCAE version 5.0.

OTHER OUTCOMES:
Expression of PDL1 | six months
  This is the description of the rate of patients with positive expression of the marker over the study population.
Expression of Nectin-4 | six months
  This is the description of the rate of patients with positive expression of the marker over the study population.
Expression of Trop-2 | six months
  This is the description of the rate of patients with positive expression of the marker over the study population.
Expression of Her-2 | six months
  This is the description of the rate of patients with positive expression of the marker over the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No